CLINICAL TRIAL: NCT05191433
Title: Effects of Mechanical Ventilation on the Diaphragm in COVID-19 Intensive Care Patients. A Post-mortem Pathology Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Professor in Anesthesia and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: COVID DIAPHRAGM
Record Dates: First submitted 2022-01-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Diaphragm Injury; Pathology; COVID-19 Acute Respiratory Distress Syndrome; Ventilation Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diaphragm is the fundamental muscle of the respiratory system. The diaphragmatic dysfunction is present in 60% of critical patients at hospital admission and up to 80% after prolonged mechanical ventilation and difficult weaning.

Risk factors associated with diaphragm dysfunction and atrophy are sepsis, trauma, sedatives, steroids, and muscle relaxants.

The main pathology characteristics of diaphragm biopsies of mechanically ventilated patients are atrophy and a reduction in contractility, determining an impact on the clinical outcome.

Shi et al. found a higher section area of the diaphragm muscle fiber in biopsies of post mortem COVID-19 patients versus negative patients, independently from days of mechanical ventilation.

The hypothesis of our study is to identify different clusters of pathological presentation in post-mortem COVID-19 mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* patients deceased in the intensive care unit positive to SARS-CoV-2 and mechanically ventilated
* post-mortem examination of the diaphragm

Exclusion Criteria:

* patients with a terminal disease and a prognosis of less than 48 hours at admission.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Deceased COVID-19 patients admitted to the intensive care unit and mechanically ventilated.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics | One week post mortem
  Evaluate if there are specific clusters in the study population and find different clinical characteristics.
Blood test characteristics | One week post mortem
  Evaluate if there are specific clusters in the study population and find different blood test characteristics.
Pathology characteristics | One week post mortem
  Evaluate if there are specific clusters in the study population and find different pathology characteristics.

SECONDARY OUTCOMES:
Mechanical ventilation | One week post mortem
  Verify if there are correlations between the clusters characteristics and the other variables in the study population mechanical ventilation.
Therapy | One week post mortem
  Verify if there are correlations between the clusters characteristics and therapy in the study population.
Arterial blood gas analysis | One week post mortem
  Verify if there are correlations between the clusters characteristics and arterial blood gas in the study population.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine
  - Azienda ospedaliero universitaria Friuli Centrale, Clinica di Anestesia e Rianimazione, Udine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCool FD, Manzoor K, Minami T. Disorders of the Diaphragm. Clin Chest Med. 2018 Jun;39(2):345-360. doi: 10.1016/j.ccm.2018.01.012. PMID 29779594
- [Background] Supinski GS, Morris PE, Dhar S, Callahan LA. Diaphragm Dysfunction in Critical Illness. Chest. 2018 Apr;153(4):1040-1051. doi: 10.1016/j.chest.2017.08.1157. Epub 2017 Sep 5. PMID 28887062
- [Background] Dres M, Goligher EC, Heunks LMA, Brochard LJ. Critical illness-associated diaphragm weakness. Intensive Care Med. 2017 Oct;43(10):1441-1452. doi: 10.1007/s00134-017-4928-4. Epub 2017 Sep 15. PMID 28917004
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Hooijman PE, Beishuizen A, Witt CC, de Waard MC, Girbes AR, Spoelstra-de Man AM, Niessen HW, Manders E, van Hees HW, van den Brom CE, Silderhuis V, Lawlor MW, Labeit S, Stienen GJ, Hartemink KJ, Paul MA, Heunks LM, Ottenheijm CA. Diaphragm muscle fiber weakness and ubiquitin-proteasome activation in critically ill patients. Am J Respir Crit Care Med. 2015 May 15;191(10):1126-38. doi: 10.1164/rccm.201412-2214OC. PMID 25760684
- [Background] Shi Z, Bogaards SJP, Conijn S, Onderwater Y, Espinosa P, Bink DI, van den Berg M, van de Locht M, Bugiani M, van der Hoeven H, Boon RA, Heunks L, Ottenheijm CAC. COVID-19 is associated with distinct myopathic features in the diaphragm of critically ill patients. BMJ Open Respir Res. 2021 Sep;8(1):e001052. doi: 10.1136/bmjresp-2021-001052. PMID 34544735